CLINICAL TRIAL: NCT03456739
Title: The Microbiome Variability and Antibiotic Resistance of Chronic Suppurative Otitis Media in Pediatric Patients in Northern Israel
Brief Title: The Microbiome Variability and Antibiotic Resistance of Chronic Suppurative Otitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0019-18-ZIV
Record Dates: First submitted 2018-02-28; First posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Suppurative Otitis Media
MeSH Terms: conditions — Otitis Media, Suppurative

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — collection of ear effusion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- suppurative otitis media with effusion
- non suppurative otitis media with effusion

SUMMARY:
ear swabs will be collected from 120 patients with established CSOM at the ear-nose-throat (ENT) outpatient clinic at the Ziv medical center, and 120 swabs will be taken from children with Otitis Media with Effusion (OME) undergoing elective tympanostomy tube insertion, serving as a control group. Ear swabs will be frozen at -80C until analysis.DNA will be purified from ear swabs, and amplified by PCR so that a barcoded 16S rRNA library from each subject will be generated. Using correlation analysis, we will compare between microbial compositions in chronic otorrhea patients vs. control groups.An additional ear swab will be collected from patients and cultured to test antibiotic resistance.

ELIGIBILITY:
Inclusion otitis media with effusion,parental informed consent, age between 1 - 9 years, no known immune deficient disorder -

Exclusion Criteria:no parental consent, known immune disorder, current acute otitis media.

-

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric patients with suppurative otitis media with effusion
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2018-04-20 (Estimated); Primary Completion 2019-04-20 (Estimated); Study Completion 2020-02-20 (Estimated)

PRIMARY OUTCOMES:
microbiome variability | 2 years
  detection of microbiome differces between suppurative and non-suppurative otitis media in pediatric patients

CONTACTS AND LOCATIONS:
Overall Officials: saqer massuod, MD, Principal Investigator — Ziv Medical Center